CLINICAL TRIAL: NCT01114750
Title: A Placebo-controlled Study of Insulin Absorption in Healthy Volunteers After Single-dose Oral Administration of Insulin in Dextran Matrix
Brief Title: A Study to Determine the Absorption of Peroral Insulin in Dextran Matrix (ORA3)
Acronym: ORA3
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Bows Pharmaceuticals AG (Industry)
Responsible Party: Nabil Al-Tawil, Karolinska Trial Alliance
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ORA3-2010-019098-14
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus
Keywords: blood glucose; blood insulin; dextran; diabetes; hyperglycemia; hypoglycemia; oral delivery; portal delivery
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Insulin in Dextran Matrix (Active Comparator): A group consisting of male healthy volunteers will be given placebo and one single dose of insulin in dextran matrix, for estimation of post-dose relative bioavailability.
  Interventions: Drug: Insulin in dextran matrix capsule (and placebo)
- Placebo (Placebo Comparator): A group consisting of male healthy volunteers will be given placebo and one single dose of insulin in dextran matrix, for estimation of post-dose relative bioavailability.
  Interventions: Drug: Insulin in dextran matrix capsule (and placebo)

INTERVENTIONS:
Drug: Insulin in dextran matrix capsule (and placebo) — Single dose capsule (and placebo)

SUMMARY:
A pharmacokinetic study on the absorption of perorally delivered insulin in dextran matrix after single dose administration.

DETAILED DESCRIPTION:
The study is a single blind, cross over study where each subject will receive a a single active dose (200 IU) of insulin in dextran matrix and placebo on two different experimental days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, age 18-40 years.
* Fasting blood glucose within the range 4.0-6.0 mmol/L at Screening, and on Day 1 before dosing ≥ 4 mmol/L. However, the subject should not be excluded from the study if the blood glucose is out of this range once the treatment period has started.
* Body Mass Index (BMI) of 20-27 kg/m2
* Medically stable as determined by history and physical examination, including vital signs.
* Screening laboratory tests must be within normal range or judged as not clinically significant by Principal investigator/Subinvestigator.
* Negative urine ketoacidosis test
* ECG including QTcB shows no clinically significant abnormality or acute ischemia
* Supine BP ≤ 139/89 mm Hg diastolic/systolic, or at the discretion of the investigator
* Able to adhere to the study visit schedule, and to understand and comply with other protocol requirements.
* Capable of giving informed consent, which must be obtained prior to any screening procedures.
* Negative laboratory screen for Hepatitis B (HBsAg and anti-HBc antibodies), Hepatitis C (anti HCV) and HIV (1&2).
* Willing to refrain from consuming alcohol 48 hours prior to dosing and throughout the period of sample collection.
* Not on any prohibited medication (See section 8.9), or at the discretion of the investigator.

Exclusion Criteria:

* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease, or any other condition which increases risk of participation in this trial in the opinion of the investigator.
* Currently known malignancy or a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been excised more than one year ago with no evidence of recurrence
* A chronic or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection (bronchiectasis), sinusitis, recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), open skin wound, or ulcer.
* Other medical conditions, drug treatments or significant medical problems that would preclude participation in a clinical trial that, in the opinion of the investigator, disqualifies the subject.
* Participation in a clinical trial within the prior 3 months
* History of GI surgery (other than appendectomy) or known GI motility disorders.
* History of a serious infection, including but not limited to hepatitis, pneumonia, or pyelonephritis, or have been hospitalized or received intravenous antibiotics for an infection, during the previous two months.
* A recent adult history of clinically significant allergic reaction to any drug.
* History of polyps in the gastrointestinal tract.
* Known to have had a substance abuse (drug or alcohol) problem within the previous 5 years
* Alcohol use within 48 hours prior to visits to the study unit.
* Unable to undergo venipunctures for study purposes because of poor tolerability or lack of easy access.
* Engaging in any strenuous exercise (such as running or weight lifting or playing any team sports such as soccer) within 48 hours prior to visits to the study unit.
* Donation of plasma within 7 days prior to the first dose.
* Donation of blood within 3 months prior to the first dose
* Difficulty in swallowing capsules.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic variable: insulin | 3-5 hours
  Estimation of insulin AUC and Cmax post dose-administration

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Al-Tawil, M.D.; Ph.D., Principal Investigator — Karolinska Trial Alliance, Stockholm
Locations (1):
- Karolinska Trial Alliance (KTA), Phase I Unit, Stockholm, Stockholm County, Sweden